CLINICAL TRIAL: NCT04872946
Title: Topical and Oral Regimen for Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Arbonne (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 008
Record Dates: First submitted 2020-10-09; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Skin Abnormalities
Keywords: skin; dermatology
MeSH Terms: conditions — Skin Abnormalities | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- InnerCalm+skin care (Experimental): An oral supplement and topical agent will be assigned.
  Interventions: Dietary Supplement: Tea; Other: Serum; Other: Moisturizer
- InnerCalm only (Experimental): An oral supplement will be assigned.
  Interventions: Dietary Supplement: Tea
- Skincare Only (Experimental): A topical agent only will be assigned.
  Interventions: Other: Serum; Other: Moisturizer

INTERVENTIONS:
Dietary Supplement: Tea — Ashwagandha(Withania somnifera) root and leaf extract (32% Withania Oligosaccharides, 10% Withanolide Glycosides, 0.5% Withaferin A) 125 mg Saffron(Crocus Sativus) stigmas extract (3.48% Crocin and 0.03% Safranal) 28mg
  Arms: InnerCalm only; InnerCalm+skin care
Other: Serum — Aqua/Water/Eau, Glycerin, Propanediol, Diheptyl Succinate, Caprylic/Capric Triglyceride, Lactococcus Ferment Lysate, Sorbitol, Dimethicone, Steareth-21, Octyldodecyl Neopentanoate, Sodium Polyacrylate, Steareth-2, Caprylyl Glycol, Hydrogenated Polydecene, Trideceth-6, Octyldodecanol, Panthenol, Sodium PCA, Azelaic Acid, Bisabolol, Capryloyl Glycerin/Sebacic Acid Copolymer, Centella Asiatica Leaf Extract, Agastache Mexicana Flower/Leaf/Stem Extract, Caprylhydroxamic Acid, Phytic Acid, Aminomethyl Propanol, Lactic Acid, Sodium Chloride, Phenoxyethanol, Sodium Benzoate.
  Arms: InnerCalm+skin care; Skincare Only
Other: Moisturizer — Aqua/Water/Eau, Glycerin, Diisopropyl Dimer Dilinoleate, Coco-Caprylate, Lactococcus Ferment Lysate, Myristyl Myristate, Dimethicone, Propanediol, Behenyl Alcohol, Glyceryl Stearate SE, Potassium Cetyl Phosphate, Palmitic Acid, Ammonium Acryloyldimethyltaurate/Beheneth-25 Methacrylate Crosspolymer, Myristyl Laurate, Caprylyl Glycol, Hydroxyethylcellulose, Myristic Acid, Tocopherol, Ethylhexylglycerin, Centella Asiatica Leaf Extract, Agastache Mexicana Flower/Leaf/Stem Extract, Helianthus Annuus (Sunflower) Seed Oil, Trisodium Ethylenediamine Disuccinate, Lactic Acid, Sodium Hydroxide, Sodium Phosphate, Disodium Phosphate, Sodium Chloride, t-Butyl Alcohol, Phenoxyethanol, Sodium Benzoate.
  Arms: InnerCalm+skin care; Skincare Only

SUMMARY:
The overall objective of this study is to assess how oral supplementation with Inner Calm and the use of topical Super Calm can affect the appearance of skin and inner wellness, such as redness, skin sensitivity, and reactionary skin.

DETAILED DESCRIPTION:
The landscape for skin health has expanded past a focused use of topicals to incorporate the use of supplementation. Notable examples include the ingestion of carotenoids and beta-carotene to augment skin antioxidant status or the role of diet on different skin conditions. The role of this investigation is to define how Inner Calm (oral supplementation) may promote healthier skin and how this may work in synergy with Super Calm (topical supplementation).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-55
* Fitzpatrick skin type 1-4
* Self-perception as sensitive skin

Exclusion Criteria:

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant or breast-feeding women
* Prisoners
* Those who have used isotretinoin in the last 6 months
* Those who have used products containing salicylic acid, beta hydroxyl acids or vitamins A, C, or E or topical retinoids or topical depigmenting agents (such as hydroquinone, kojic acid, azelaic acid, or others in opinion of the investigator) in the last 14 days
* Those who are currently smoking or have smoked within the past 3 years.
* Those who have had a recent surgical or cosmetic procedure in the last 3 months that can affect facial wrinkles, redness, or hyperpigmentation, such as botulinum toxin injections, chemical peels, laser-based therapies to the face, or face lift surgeries
* Subjects with known allergy to any of the components of Inner Calm or Skin Calm
* Those that are unwilling to discontinue use of any other nutritional supplements including antioxidants, herbs, or protein-based supplements for 2 weeks prior to and during their participation.
* Subjects with a diagnosis of acne

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Changes in appearance of facial redness | 8 weeks
  Photographic image analysis
Changes in appearance of facial pigmentation | 8 weeks
  Photographic image analysis

SECONDARY OUTCOMES:
Changes in appearance of facial redness before and after treatment | 8 weeks
  SkinColorCatch colorimeter RGB range: 25-246 per channel
Subjective report of skin reactivity | 8 weeks
  Topical Clinical Questionnaire
Subjective report of sleep quality and quantity | 8 weeks
  Pittsburg Sleep Quality Index survey (PSQI)
Subjective report of mood and energy | 8 weeks
  Abbreviated Profile of Mood States Survey (POMS)
Subjective report of calmness of mind | 8 weeks
  Inner and Outer Calm Questionnaire
Subjective report of calmness of skin | 8 weeks
  Inner and Outer Calm Questionnaire
Changes in appearance of facial redness | 4 weeks
  Photographic image analysis
Changes in appearance of facial pigmentation | 4 weeks
  Photographic image analysis

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — Integrative Skin Science and Research Institute
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States